CLINICAL TRIAL: NCT00565032
Title: Postpartum Thyroid Measures and Mood
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Other Study IDs: 9899015
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; thyroxine; thyroid antibodies; thyroid stimulating hormone; Edinburgh Postnatal Depression Scale (EPDS)
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Women with abnormal serum thyroid antibody levels or abnormal TSH and/or T4 values are more likely than their normal counterparts to have higher scores on a common postpartum depression screening test.

DETAILED DESCRIPTION:
This small pilot study was an attempt to corroborate a relationship between quantified mood and thyroid measures, using the numerical scores obtained from a common depression screen, the Edinburgh Postnatal Depression Scale (EPDS), as a continuum. Mood scores were compared with presence of thyroid autoantibodies and plasma concentrations of free T4 and TSH.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* In third trimester of pregnancy when recruited
* Negative for the following drugs detected by a urine drug screen:

  * Amphetamines
  * Barbiturates
  * Benzodiazepines
  * Cocaine
  * Opiates
  * Phencyclidine metabolites (PCP), and tricyclic antidepressants
  * Vaginal delivery
  * Screened negative for major depressive disorder on the Edinburgh Postnatal Depression Scale (EPDS) at her prenatal enrollment in the study
  * Receiving a score of 12 or lower out of a possible 30

Exclusion Criteria:

* Under age 18
* Positive for any of the following drugs:

  * Amphetamines
  * Barbiturates
  * Benzodiazepines
  * Cocaine
  * Opiates
  * Phencyclidine metabolites (PCP), and tricyclic antidepressants
  * Cesarean delivery
  * EPDS score over 12 at prenatal screening test

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects were patients from two Oklahoma State University Center for Health Sciences (OSUCHS) clinics in Tulsa, Oklahoma.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2000-01; Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Numerical score on the Edinburgh Postnatal Depression Scale | seven weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary H. Watson, PhD, Study Director — Philadelphia College of Osteopathic Medicine Georgia Campus
Locations (1):
- Oklahoma State University Center for Health Sciences Houston Park Obstetrics Clinic, Tulsa, Oklahoma, United States

REFERENCES:
- [Derived] McCoy SJ, Beal JM, Payton ME, Stewart AL, DeMers AM, Watson GH. Postpartum thyroid measures and depressive symptomology: a pilot study. J Am Osteopath Assoc. 2008 Sep;108(9):503-7. PMID 18806079